CLINICAL TRIAL: NCT06936410
Title: Intraoperative Infusion of Lidocaine vs. Dexmedetomidine for Decreasing Tourniquet Induced Hypertension (TIH) in Ambulatory Arthroscopic Knee Surgeries Under General Anesthesia
Brief Title: Using Lidocaine or Dexmedetomidine to Help Control Blood Pressure Spikes From a Tourniquet During Knee Surgery
Acronym: torniquet
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa mahmoud bahaa eldin mohamed taha, lecturer of anaesthesia , surgical ICU and pain -cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-76-2023
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Tourniquet Hypertension
Keywords: lidocaine; dexmedetomidine
MeSH Terms: interventions — Lidocaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lidocaine group (group L) (Active Comparator): patients received Lidocaine 2%, 1 mg/kg, IV bolus over 10 mins after the induction of anaesthesia , followed by Lidocaine infusion (2 mg/kg/h) diluted in 50 ml of normal saline with a maximum dose of 200 mg/h. The tourniquet was inflated 10 minutes after the start of the Lidocaine infusion then the Lidocaine infusion stopped at the time of tourniquet deflation
  Interventions: Drug: Dexmedetomidine HCL Injection
- dexmedetomidine group (group D) (Active Comparator): atients received a loading dose of Dexmedetomidine-Pfizer (0.8 μg·kg-1 over 10 min) followed by continuous infusion of Dexmedetomidine (0.4 μg·kg-1.h-1) diluted in 50 ml of normal saline. The tourniquet was inflated 10 mins after the start of Dexmedetomidine infusion then the Dexmedetomidine infusion stopped at the time of the tourniquet deflation.
  Interventions: Drug: Lidocaine 2% Injectable Solution

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — patients received Lidocaine 2%, 1 mg/kg, IV bolus over 10 mins after the induction of anaesthesia , followed by Lidocaine infusion (2 mg/kg/h) diluted in 50 ml of normal saline with a maximum dose of 200 mg/h. The tourniquet was inflated 10 minutes after the start of the Lidocaine infusion then the Lidocaine infusion stopped at the time of tourniquet deflation
  Arms: dexmedetomidine group (group D)
Drug: Dexmedetomidine HCL Injection — patients received a loading dose of Dexmedetomidine-Pfizer (0.8 μg·kg-1 over 10 min) followed by continuous infusion of Dexmedetomidine (0.4 μg·kg-1.h-1) diluted in 50 ml of normal saline. The tourniquet was inflated 10 mins after the start of Dexmedetomidine infusion then the Dexmedetomidine infusion stopped at the time of the tourniquet deflation.
  Arms: lidocaine group (group L)

SUMMARY:
Knee pain is very common, and more people are having minor knee surgeries done through a small camera (arthroscopy), often as outpatients. During these surgeries, a device called a tourniquet is used to reduce bleeding by stopping blood flow to the leg. However, this can sometimes cause a sharp rise in blood pressure-a condition known as tourniquet-induced hypertension (TIH), which happens in about 67% of patients under general anesthesia.

this study looked at two different drugs-Dexmedetomidine and Lidocaine- to see which one works better in preventing this blood pressure rise during surgery.

Dexmedetomidine is a medicine that calms the nervous system and helps lower blood pressure and pain, but it can sometimes cause side effects like a slow heart rate and low blood pressure. Lidocaine, commonly used to numb pain, also helps with inflammation and controlling pain sensitivity.

In this study, both drugs helped reduce TIH, but Dexmedetomidine was more effective. However, it came with more side effects compared to Lidocaine.

DETAILED DESCRIPTION:
Knee pain is very common and ambulatory knee arthroscopic surgery has increased significantly. Clinical studies comparing spinal anaesthesia to general anaesthesia (GA), have found that GA resulted in slightly shorter hospital stay, earlier mobilization, and fewer cases of urinary retention; that is why the investigators preferred in this study to choose the general anaesthesia over spinal anaesthesia in patients undergoing ambulatory knee arthroscopic surgeries.

Tourniquet induced hypertension defined as an increase of at least 30% in the systolic blood pressure or diastolic blood pressure within one hour of the tourniquet inflation, which may affect the response to analgesia and the need for antihypertensive drug. The incidence of TIH in patients undergoing general anaesthesia using tourniquet is 67%.

Previous studies were conducted to investigate the effect of different drugs such as Lidocaine, Ketamine or Dexmedetomidine in managing TIH.

This study used Dexmedetomidine to decrease the TIH, and another one, used Lidocaine as bolus plus infusion to decrease the TIH, but to our knowledge no study was done to compare between both drugs in decreasing TIH. Dexmedetomidine is a selective, short acting agonist of the alpha 2 receptors, it has a sympatholytic effect, in addition to antihypertensive, anxiolytic, sedative and analgesic effects.

Lidocaine is an anti-inflammatory drug with an analgesic and anti-hyperalgesia effect. It is also used in attenuating the stress response that can occur while using the laryngoscope.

This study aimed to compare the effect of IV infusion of dexmedetomidine with the effect of IV Lidocaine in decreasing the TIH in patients undergoing ambulatory arthroscopic knee surgeries using the tourniquet under general anaesthesia.

This randomized, comparative and double blinded study on 180 patients undergoing ambulatory knee arthroscopy under general anaesthesia using tourniquet. Patients were randomly allocated into two equal groups: Lidocaine group (group L): patients received lidocaine 2%, 1 mg/kg and dexmedetomidine group (group D): patients received a loading dose of (0.8 μg·kg-1 over 10 min) followed by continuous infusion of (0.4 μg·kg-1.h-1) diluted in 50 ml of normal saline.

ELIGIBILITY:
Inclusion Criteria:

Patients (males and females) of ASA class I or II, age from 18-60 years old, undergoing ambulatory knee arthroscopy under general anaesthesia using tourniquet.

Exclusion Criteria:

1. Patients with uncontrolled systemic diseases (e.g., diabetes mellitus, hypertension, and chronic obstructive lung disease),
2. Patients with significant organ dysfunctions (e.g., cardiac, respiratory, renal, or liver disorders).
3. Patients with morbid obesity (BMI >35).
4. Patients with a history of allergy to the drugs used in this study.
5. Patients who have history of chronic use of opioids.
6. Cases with tourniquet times of less than 60 minutes or longer than 150 minutes were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of tourniquet induced hypertension | from 60 minutes after tourniquet inflation till end of surgery
  which is defined as increase in the SBP or DBP 30% from the baseline reading in both groups, at 60 mins after tourniquet inflation

SECONDARY OUTCOMES:
Hemodynamic measurements: SBP, DBP, MAP and HR. | from baseline till 1 hour after end of operation

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes